CLINICAL TRIAL: NCT06841081
Title: Super-Supporters - Specially Trained Staff to Facilitate Virtual Care for Vulnerable Patients and Family Caregivers: A Real-world Implementation and Evaluation Across North and South Carolina
Brief Title: Super-Supporters - Virtual Care Technology Navigators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB00078662
Record Dates: First submitted 2025-02-14; First posted 2025-02-24 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-05

CONDITIONS: Telemedicine
Keywords: virtual health; virtual telehealth; telemedicine

STUDY DESIGN:
Intervention Model Description: The study design is a randomized implementation of the quality improvement program, the "Super-Supporter" program, with post-implementation evaluation using patient assessments (24 hour survey and six month survey). Investigators will use a randomization protocol especially suited to comparison of a best standard compared with an enhanced intervention: the Zelen protocol. In this protocol, randomization occurs prior to calling patients and enrolling them in the evaluation. A cluster-randomized design will be used with 1-week intervals as the randomization cluster. All patients called within a given week will be randomized to the same group. Allocation of weeks to group will be determined by a block-randomization table establish prior to trial initiation.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (Active Comparator): At the beginning of the call for patients randomized to Enhanced Usual Care, the Super Supporter will identify themselves, verify they are speaking with the patient, confirm the patient has an upcoming video visit, and ask if they are prepared to log into the video visit. If they are not, the Super Supporter will offer to send written instructions to the patient and refer the patient to their clinical team if they have unresolved issues. Then, they will tell the patient about the research the team is conducting and ask if they would like to participate. If so, the Super Supporter will follow the same protocol for Super Supporter intervention in telling them about the study. If they are interested, as with the other randomized group, REDCap will send the survey by email link with the info sheet included at the beginning.
  Interventions: Other: Enhanced Usual Care
- Super Supporter Support (Experimental): At the beginning of the call for patients randomized to Super Supporter support, the Super Supporter will identify themselves, verify they are speaking with the patient, confirm the patient has an upcoming video visit, and ask if they would like assistance connecting with their upcoming visit. Once the Super Supporter has assisted and trouble shot with the patient and conducted a practice video visit, they will tell the patient about the opportunity to participate in the research study and ask if they would like to participate . If so, the Super Supporter will select yes that they are interested in REDCap and REDCap will automatically send the initial survey with the verbal consent included as the face page to the survey.
  Interventions: Other: Super Supporter Support

INTERVENTIONS:
Other: Enhanced Usual Care — Offer written instructions to the patient and refer the patient to their clinical team if they have unresolved issues.
  Arms: Enhanced Usual Care
Other: Super Supporter Support — Assist and troubleshoot with the patient including a practice video visit.
  Arms: Super Supporter Support

SUMMARY:
The Super-Supporter Program is designed to provide pre-visit support to patients who are at risk of not being able to participate in Virtual Care modalities (specifically, Clinical Video Visits). Patient technology navigators (Super-Supporters) will reach out before video visits and help the patient connect more easily and successfully with their providers in Virtual Care appointments.

DETAILED DESCRIPTION:
The Super Supporter Technology Navigator Program was designed to support patients, across the health system, to connect more easily and successfully with their providers in Virtual Care appointments. Super Supporters call patients in advance of Virtual Care appointments to remind them of their appointment, ensure that they have a device on which to conduct the appointment, set up the device for a successful Virtual Care appointment, help them set up and log into their patient portal account, and practice connecting with their provider using a practice virtual video visit. This research study is designed to determine differences in connection rate, patient reported health, patient access and responses to a healthcare climate questionnaire by comparing those helped by a Super Supporter and those supported by an Enhanced Usual Care program.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a video visit with a provider at Atrium Health (all locations)
* Identified as at risk of a failed video visit using criteria (1) a failed prior video visit (a discrete data field noting a prior visit was unsuccessful or converted to telephone-only visit), or 2) no prior access to the Electronic Health Record-connected patient portal

Exclusion Criteria:

* Patient plans to change visit to in-person or telephone only
* Patient declines assistance from the Super-Supporter program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1111 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Rate of Successful Video Visits | Up to Week 3
  Data will be collected from electronic health record review

SECONDARY OUTCOMES:
Health Care Climate Questionnaire (HCCQ) | Month 6
  This 15-item scale assesses participants' perceptions of the degree of autonomy support versus controllingness of relevant healthcare providers. Total score range is 15-105 with higher scores indicating a more positive perception of healthcare communication.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Houston, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Atrium Health, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No
This project by a specific endowment and thus does not have a sharing requirement.

DOCUMENTS (1):
  • Informed Consent Form (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT06841081/ICF_000.pdf